CLINICAL TRIAL: NCT04178512
Title: Effect of Intrathecal Dexamethasone Versus Fentanyl on Post Spinal Shivering in Patients Undergoing Transurethral Prostatectomy
Brief Title: Intrathecal Additives to Prevent Post Spinal Shivering in Transurethral Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Fatma Mahmoud Ahmed, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: transurethral prostatectomy
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group Dexamethasone (Active Comparator): Patients will receive 8 mg of dexamethasone(2ml) in addition to 2ml of hyperbaric bupivacaine 0.5% (total volume 4 ml) intrathecal injection.
  Interventions: Drug: Drug:dexamethasone in group Dexamethasone,fentanyl in group Fentanyl,normal saline 0.9%in group Control
- group Fentanyl (Active Comparator): patients will receive 20 microgram fentanyl(diluted in sterile normal saline0.9% to 2ml)in addition to 2ml of hyperbaric bupivacaine 0.5%(total volume 4 ml) intrathecal injection.
  Interventions: Drug: Drug:dexamethasone in group Dexamethasone,fentanyl in group Fentanyl,normal saline 0.9%in group Control
- group Control (Active Comparator): patients will receive 2ml of sterile normal saline0.9% in addition to 2ml of hyperbaric bupivacaine o.5% (total volume 4 ml) intrathecal injection.
  Interventions: Drug: Drug:dexamethasone in group Dexamethasone,fentanyl in group Fentanyl,normal saline 0.9%in group Control

INTERVENTIONS:
Drug: Drug:dexamethasone in group Dexamethasone,fentanyl in group Fentanyl,normal saline 0.9%in group Control — prevention of shivering after spinal anesthesia in patients undergoing trans urethral prostatectomy through injection of spinal additives
  Other Names: Intrathecal additives

SUMMARY:
Spinal anesthesia is the technique of choice in transurethral prostatectomy.However,one of the common complications of spinal anesthesia is shivering which is even exaggerated in patients undergoing transurethral prostatectomy.this high incidence is most probably caused by sympathetic block and use of large amount of irrigation fluid during surgery.There are two methods to reduce shivering.Previous studies showed that intrathecal fentanyl is an appropriate method to reduce shivering.Intrathecal dexamethasone could reduce shivering by regulating immune responses.

DETAILED DESCRIPTION:
Shivering is an involuntary repetitive contractions of skeletal muscles that increases the basal metabolism and is considered to be a defense mechanism for regulating body temperature in adults .

Post spinal shivering may cause discomfort to the patient,and may aggravate wound pain by stretching incisions and increases intracranial and intra ocular pressure.Shivering may increase tissue oxygen demand as much as 500% and is accompanied by increase in minute ventilation and cardiac output to maintain aerobic metabolism.

Tympanic temperature will be recorded preoperatively,after establishment of spinal anesthesia,and every 15 minutes til the end of operation.Core temperature below 36.5 C is considered as hypothermia Shivering intensity will be assessed with a five -point scale validated by Crossly and Maharaj.

Adverse events like hypotension,bradycardia, respiratory depression,nausea and vomiting will be recorded and treated.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American society of anesthesiologists) physical status grade I-II
* BMI(body mass index) less than 35 kg/m2
* patients undergoing transurethral prostatectomy

Exclusion Criteria:

* patient refusal.
* patients with contraindications to spinal anesthesia e.g coagulopathy,anti coagulant therapy,allergy to local anesthetic,psychological disorders,...
* patient with advanced cardiopulmonary diseases or thyroid diseases.
* patients on corticosteroids therapy or on Alpha2 blocker orAlcohol.
* patients with initial body temperature above 37.5 C or below 36.5 C.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
incidence of shivering | intraoperative every 15 min till the end of surgery and in the recovery room for 2 hours
  compare between the effect of intrathecal dexamethasone and intrathecal fentanyl on the incidence of shivering in patients undergoing transurethral prostatectomy

SECONDARY OUTCOMES:
comparative assessment between both drugs | intraoperative and in the recovery room for 2 hours
  compare between both drugs as regards severity of shivering,hypothermia,hemodynamic changes and side effects of the used drugs

CONTACTS AND LOCATIONS:
Overall Officials: Abeer HM Elsawy, MD, Study Chair — Faculty of medicine,Zagazig University,Egypt